CLINICAL TRIAL: NCT01064011
Title: A Prospective Randomized, Controlled Trial for Treatment of Intraventricular Hemorrhage: External Ventricular Drainage and Intraventricular Thrombolysis vs. External Ventricular Drainage and Endoscopic Evacuation
Brief Title: Prospective Randomized, Controlled Trial for Treatment of Intraventricular Hemorrhage
Acronym: IVH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Yu-hung Kuo, MD, Albany Medical College
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-01

CONDITIONS: Intraventricular Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- External Ventricular drainage, Intraventricular Thrombolysis (Other)
  Interventions: Procedure: Rt-PA thrombolysis
- External Ventricular Drainage and Endoscopic Evacuation (Other)
  Interventions: Procedure: endoscopic hematoma evacuation

INTERVENTIONS:
Procedure: Rt-PA thrombolysis — patients will be administered a total of six doses of rt-PA (each 1 mg/ml) through the external ventricular drain every eight hours.
  Arms: External Ventricular drainage, Intraventricular Thrombolysis
Procedure: endoscopic hematoma evacuation — In the operating room under general anesthesia, the external ventricular drain will be removed and the burr hole enlarged to allow for entry of the endoscope. The neuroscope will be introduced through the burr hole down the prior external ventricular drain tract into the ipsilateral ventricle. utilizing a standard technique combining gentle aspiration, continuous irrigation, and grasping forceps,the intraventricular hematoma will be evacuated. After the evacuation the endoscope will be removed and an external ventricular drain will be reattached to a closed system and permitted to drain post-operatively.
  Arms: External Ventricular Drainage and Endoscopic Evacuation

SUMMARY:
Intraventricular hemorrhage comprises about 15% of the 500,000 strokes that occur annually in the United States. In the emergent setting, patients with obstructive hydrocephalus are routinely treated with placement of an external ventricular drain. This study will compare the effect of external ventricular drainage plus intraventricular thrombolysis versus external ventricular drainage plus endoscopic evacuation on neurologic outcomes for patients with hydrocephalus from intraventricular hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Radiographic evidence of intraventricular hemorrhage with hydrocephalus
* Admission Glasgow Coma Scale ≥ 5 (motor score ≥ 2)
* Placement of an external ventricular drain with an opening pressure >20 mm Hg

Exclusion Criteria:

* Intraventricular hemorrhage secondary to cerebral aneurysm, arteriovenous malformation, or tumor
* Coagulopathy (Platelet count <100,000, International normalized ratio >1.5. Reversal of warfarin is permitted.)
* Age <18 or >75
* Pregnancy (positive pregnancy test)
* Clotting disorders
* Medical contraindications to administration of general anesthesia as determined by the attending anesthesiologist
* Medical contraindications to surgery as determined by the attending neurosurgeon
* Contraindication to recombinant tissue plasminogen activator administration:

  * Evidence of enlargening intracranial hemorrhage as evidenced by an increase in intracranial hemorrhage volume (>5 ml) on CT obtained after EVD placement
  * Internal bleeding, involving retroperitoneal sites, or the gastrointestinal, genitourinary, or respiratory tracts
  * Superficial or surface bleeding, observed at vascular puncture and access sites (e.g. venous cutdowns, arterial punctures) or site of recent surgical intervention
* Evidence of cerebrospinal infection by Gram stain or culture
* Advanced directive indicating Do Not Resuscitate or Do Not Intubate status

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States